CLINICAL TRIAL: NCT03534466
Title: Evaluation of Long-Term Gait Development in Infants With Neonatal Encephalopathy Using Infant Treadmill
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was concluded as planned upon reaching its predetermined endpoint, which included the completion of data collection and achievement of the necessary sample size for statistical significance.
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Shanghai High-risk Infants Early Intervention Center (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHFudanU_NNICU9
Record Dates: First submitted 2018-02-22; First posted 2018-05-23 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Hypoxic-Ischemic Encephalopathy; Periventricular Leukomalacia; Intraventricular Hemorrhage Neonatal; Bilirubin Encephalopathy; Kernicterus; Hypoglycemia, Neonatal; Cerebral Infarction
Keywords: treadmill; infants; neonatal encephalopathy; neonatal brain injury
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Leukomalacia, Periventricular; Kernicterus; Hypoglycemia; Cerebral Infarction

STUDY DESIGN:
Intervention Model Description: Parallel Assignment All subjects were divided into two groups: intervention group A (treadmill intervention + routine physical rehabilitation therapy) and positive control group (receiving routine physical rehabilitation therapy only).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Baby treadmill + conventional physical rehabilitation training
  Interventions: Device: Baby treadmill; Behavioral: Conventional physical rehabilitation training
- positive control group (Active Comparator): Conventional physical rehabilitation training only
  Interventions: Behavioral: Conventional physical rehabilitation training

INTERVENTIONS:
Device: Baby treadmill — The newborns who received treadmill intervention were stimulated by running 3 times a week for a total of 10 minutes each time (complete in 5 cycles, 2 minutes per cycle, 2 minutes after the completion of one cycle and rest for 2 minutes to start the next cycle). Until the completion and completion of the five cycles). During the remaining four days of each week, other physical rehabilitation training is carried out by the rehabilitator in accordance with the established rehabilitation plan. The stimulation of running lasted from 3 months of corrected gestational age to being able to walk alone for 3 steps or to correct for 18 months.
  Arms: intervention group
Behavioral: Conventional physical rehabilitation training — Suitable for general physical rehabilitation training of all infants with cerebral palsy.

SUMMARY:
There have been many studies on the use of running training in older children to improve gait development in children with cerebral palsy. The aim of our study was to conduct early treadmill training in infants who were highly suspected of cerebral palsy and to follow up on their long-term gait development.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age < 33W;
2. Correction of gestational age < 3 months;
3. It has been diagnosed as hypoxic-ischemic encephalopathy, periventricular intraventricular hemorrhage, periventricular leukomalacia, bilirubin encephalopathy, persistent hypoglycemia and cerebral infarction.
4. There was no other therapeutic intervention before entering the study;
5. Informed consent is signed by the family.

Exclusion Criteria:

1. Brain injury caused by central or peripheral infection (cerebrospinal fluid positive / torch test positive / three major conventional culture positive);
2. Brain damage caused by convulsion;
3. Metabolic brain damage caused by genetic defects;
4. Suffering from known severe congenital malformations;
5. Definite head trauma during labor or postpartum;
6. Peripheral neuromuscular disease or abnormal skeletal system.

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
step frequency | The length of time from birth to the corrected age of 18 months
  This variable is a number that records the infants' number of coordinated gaits in all gait training processes.
age of onset of independent walking | The length of time from birth to the corrected age of 2 years
  This variable is a gait parameter, recording a point in time the baby will start walking independently.

SECONDARY OUTCOMES:
age of onset of walking with assistance | The length of time from birth to the corrected age of 2 years
  This variable is a gait parameter, recording a point in time the baby will start walking with assistance.
step length | The length of time from birth to the corrected age of 18 months
  The length of displacement formed by the same foot after completing a gait.
step width | The length of time from birth to the corrected age of 18 months
  The vertical distance between the parallel lines of two medial plantar edges
gait double-limb support | The length of time from birth to the corrected age of 18 months
  The percentage of two-limb support gait in the whole training process.
gait ankle plantar flexion | The length of time from birth to the corrected age of 18 months
  The percentage of gait ankle plantar flexion in the whole training process.
toe-off | The length of time from birth to the corrected age of 18 months
  The percentage of toe-off gait in the whole training process.
gait ankle dorsiflexion | The length of time from birth to the corrected age of 18 months
  The percentage of ankle dorsiflexion gait in the whole training process.

CONTACTS AND LOCATIONS:
Locations (1):
- Children Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vasudevan EV, Patrick SK, Yang JF. Gait Transitions in Human Infants: Coping with Extremes of Treadmill Speed. PLoS One. 2016 Feb 1;11(2):e0148124. doi: 10.1371/journal.pone.0148124. eCollection 2016. PMID 26828941
- [Result] Teulier C, Lee DK, Ulrich BD. Early gait development in human infants: Plasticity and clinical applications. Dev Psychobiol. 2015 May;57(4):447-58. doi: 10.1002/dev.21291. Epub 2015 Mar 18. PMID 25782975
- [Result] Siekerman K, Barbu-Roth M, Anderson DI, Donnelly A, Goffinet F, Teulier C. Treadmill stimulation improves newborn stepping. Dev Psychobiol. 2015 Mar;57(2):247-54. doi: 10.1002/dev.21270. Epub 2015 Feb 2. PMID 25644966
- [Result] de Klerk CC, Johnson MH, Heyes CM, Southgate V. Baby steps: investigating the development of perceptual-motor couplings in infancy. Dev Sci. 2015 Mar;18(2):270-80. doi: 10.1111/desc.12226. Epub 2014 Aug 13. PMID 25123212
- [Result] Madhavan S, Campbell SK, Campise-Luther R, Gaebler-Spira D, Zawacki L, Clark A, Boynewicz K, Kale D, Bulanda M, Yu J, Sui Y, Zhou XJ. Correlation between fractional anisotropy and motor outcomes in one-year-old infants with periventricular brain injury. J Magn Reson Imaging. 2014 Apr;39(4):949-57. doi: 10.1002/jmri.24256. Epub 2013 Oct 17. PMID 24136687
- [Result] Angulo-Barroso RM, Tiernan C, Chen LC, Valentin-Gudiol M, Ulrich D. Treadmill training in moderate risk preterm infants promotes stepping quality--results of a small randomised controlled trial. Res Dev Disabil. 2013 Nov;34(11):3629-38. doi: 10.1016/j.ridd.2013.07.037. Epub 2013 Sep 4. PMID 24012586